CLINICAL TRIAL: NCT00380627
Title: Quality of Life With Arcoxia in Women With Dysmenorrhea
Brief Title: Quality of Life With Arcoxia in Women With Dysmenorrhea (0663-094)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0663-094; 2006_035
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Etoricoxib; Duration of Therapy

INTERVENTIONS:
Drug: MK0663, Arcoxia, etoricoxib / Duration of Treatment: 3 Days

SUMMARY:
Allow gynecologists to gain experience with arcoxia for treatment of dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women older than 18 years old and younger than 25 years old
* Voluntary agreement to participate in the study and signature of informed consent
* Women with clinical diagnosis of dysmenorrhea

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea due to: endometriosis, adenomyosis, malformations of Muller's conducts, uterine fibromyomas, ovarian cystic, pelvic varicocoele, inflammatory pelvic disease, adherences, intrauterine devices, cervical channel stenosis, etc.
* Patients with diagnosis of acute inflammatory abdomen
* Patients with diagnosis of congestive heart disease, stroke (1 year), unstable angina, and history of myocardial infarction
* Women auto prescribing rescue medication for dysmenorrheal pain during the study
* Women with a diagnosis of mild dysmenorrhea

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 337
Dates: Start 2005-09-01 (Actual); Primary Completion 2006-01-31 (Actual); Study Completion 2006-01-31 (Actual)

PRIMARY OUTCOMES:
Perception of menstrual pain, through the analog verbal scale during three days.

SECONDARY OUTCOMES:
Quality of life measures during three days.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC